CLINICAL TRIAL: NCT00254020
Title: The Role of Cytokine-Serotonin Interactions in Post-Stroke Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 380-2004
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: stroke; depression; cytokines; serotonin; citalopram
MeSH Terms: conditions — Depression; Stroke | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Citalopram — Patients who are found to have major depression will be referred to a psychologist
  Other Names: Celexa

SUMMARY:
Depression is a common and often serious problem occurring in stroke patients. Inflammatory hormones, known as cytokines, are stimulated by an activated immune system and sometimes become active following a stroke. They may be responsible for altering levels of key neurotransmitters and their metabolites in the blood and brain of stroke patients. The investigators' objective is to examine whether increased cytokine activity following a stroke may be the cause of an increased presence or severity of depression or cognitive impairment among stroke patients, as a result of tryptophan depletion and/or kynurenine activation. They are recruiting patients within one month of their strokes and measuring levels of key markers in their blood. Patients are assessed for the presence of depressive and/or cognitive symptoms and treated with an antidepressant if needed. The investigators expect to show that cytokine activation is related to depression and/or cognitive impairment among stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Gender: male or female
* Language: speaks and understands English
* Clinical diagnosis of stroke according to World Health Organization MONICA Project and recent (< 3 months) cerebral infarctions
* Written, informed consent
* Depressed group only: diagnosis of a major depressive episode according to the depression module of the Structured Clinical Interview for the DSM-IV (SCID-IV)

Exclusion Criteria:

* Subarachnoid hemorrhage
* Intracranial hemorrhage
* Significant acute medical illness including: drug overdose, severely disturbed liver, kidney or lung function, anemia, hypothyroidism, or uncontrolled diabetes
* Significant acute neurologic illness including: impaired consciousness, Parkinson's disease, Huntington's chorea, progressive supranuclear paralysis, brain tumor, subdural hematoma, multiple sclerosis, hydrocephalus, Binswanger's disease, or severe aphasia
* Presence of a premorbid Axis I psychiatric diagnosis (eg. schizophrenia, bipolar disorder)
* Depressed group only: contraindications to receiving treatment with citalopram (including previous nonresponse) or serious risk of suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-06; Primary Completion 2011-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Centre for Epidemiological Studies-Depression Scale (CES-D) | Baseline, 6 weeks, 12 weeks
Mini Mental State Examination (MMSE) | Baseline, 6 weeks, 12 weeks
NINCDS-CSN Vascular Cognitive Impairment Battery | Baseline, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | Baseline, 6 weeks, 12 weeks
NIH Stroke Scale | Baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - York Central Hospital, Richmond Hill, Ontario
  - St. John's Rehabilitation Hospital, Toronto, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Baycrest, Toronto, Ontario

REFERENCES:
- [Result] Bensimon K, Herrmann N, Swardfager W, Yi H, Black SE, Gao FQ, Snaiderman A, Lanctot KL. Kynurenine and depressive symptoms in a poststroke population. Neuropsychiatr Dis Treat. 2014 Sep 22;10:1827-35. doi: 10.2147/NDT.S65740. eCollection 2014. PMID 25285006